CLINICAL TRIAL: NCT06866262
Title: Phase I/II Trial of Inulin Gel in Combination With Ipilimumab and Nivolumab in Advanced Renal Cell Carcinoma [ICON Trial]
Brief Title: Inulin Gel in Combination With Ipilimumab and Nivolumab for the Treatment of Metastatic or Locally Advanced Kidney Cell Cancer, ICON Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2024.067; NCI-2025-01192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00262019 (Other: University of Michigan); UMCC 2024.067 (Other: University of Michigan Comprehensive Cancer Center); HT94252310926 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Clear Cell Renal Cell Carcinoma; Locally Advanced Sarcomatoid Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Sarcomatoid Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Biopsy; Specimen Handling; Inulin; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 5, patients receive nivolumab monotherapy IV over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study. Patients may optionally undergo biopsy during screening, on study, and at disease progression.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Other: Questionnaire Administration
- Safety run-in & Arm B (nivolumab, ipilimumab, inulin gel) (Experimental): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 5, patients receive nivolumab monotherapy IV over 30 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inulin gel PO BID for 52 weeks in the absence of disease progression or unacceptable toxicity. Patients receiving benefit from study treatment may optionally continue receiving inulin gel PO BID beyond 52 weeks at the discretion of the treating physician and in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study. Patients may optionally undergo biopsy during screening, on study, and at disease progression.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Dietary Supplement: Inulin; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Dietary Supplement: Inulin — Given PO
  Arms: Safety run-in & Arm B (nivolumab, ipilimumab, inulin gel)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I/II trial tests the safety and effectiveness of inulin gel in combination with ipilimumab and nivolumab in treating patients with kidney cell cancer (renal cell carcinoma [RCC]) that has spread from where it first started (primary site) to other places in the body (metastatic) or has spread to nearby tissue or lymph nodes (locally advanced). Inulin is a common food additive fermentable prebiotic fiber beneficial for a healthy gut microbiome. The microbiome is the collection of all microbes, such as bacteria, fungi, viruses, and their genes, that naturally live on and inside the body. Inulin may also be used for cancer prevention and heart health, but there is less evidence to support those uses. The gut microbiome profile may improve the effectiveness of drugs called immune checkpoint inhibitors, such as ipilimumab and nivolumab. Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving inulin gel in combination with ipilimumab and nivolumab may be safe and effective in treating in patients with metastatic or locally advanced RCC.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age on the day of signing informed consent.
* Candidate for ipilimumab and nivolumab therapy for metastatic renal cancer per the treating physician investigator.
* Patient has a performance status of ≤ 2 on the Zubrod performance scale.
* Patient has a histological or cytological diagnosis of renal cancer with clear cell or sarcomatoid component.
* Radiologic or clinical evidence of metastatic disease, or progressive locally advanced disease.
* Absolute neutrophil count ≥ 1,500/uL.
* Platelets ≥ 75K/μL.
* Hemoglobin ≥ 8.5 g/dL.
* Calculated creatinine clearance is ≥ 30 ml/min as per the Cockroft-Gault formula.
* Direct bilirubin ≤ 1.5 x upper limit of normal (ULN) OR total bilirubin levels ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN.
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x ULN except for patients with liver metastases, AST/ALT should be ≤ 5 x ULN.
* Patient received no prior systemic anti-cancer therapy for metastatic disease.
* Patient has evaluable or measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Bone metastases, pleural effusion or ascites will be considered evaluable disease sites.

  * Tumor mass: Must be accurately measurable in at least 1 dimension (longest diameter to be recorded) with a minimum size of:

    * 10 mm by CT scan (CT scan slice thickness no greater than 5 mm,

Or:

* 20 mm by chest X-ray (if clearly defined and surrounded by aerated lung). With or without malignant lymph nodes: ≥ 15 mm in short axis when assessed by CT scan (CT scan slice thickness must be ≤ 5 mm). The measurement should be two dimensions at axial plane. The short axis should be in perpendicular to long diameter.

  * Ability to understand and the willingness to review and sign a written informed consent.
  * Both male and female patients must agree to use adequate contraceptive measures to prevent pregnancy throughout the duration of study therapy and a minimum of -5 months after stopping therapy per package insert of ipilimumab and nivolumab.
  * Ability to ingest oral therapy.
  * Female patient of childbearing capacity has a negative pregnancy test within 7 days of starting study therapy.

Exclusion Criteria:

* The subject has received cytotoxic therapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) or immunosuppressants (excluding steroids) within 4 weeks or antibiotics within 2 weeks of starting study therapy.
* Patient is currently enrolled in another clinical trial testing another investigational agent, or concurrently in another approved systemic anti-cancer therapy for renal cancer.
* Patient is on chronic systemic steroid therapy at doses > 10 mg/day prednisone equivalent or on any other immunosuppressive therapy within 7 days prior to day 1 of therapy. Exception-Replacement steroid doses for adrenal insufficiency are permitted as necessary.
* Subjects with active and uncontrolled autoimmune disease. Subjects with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll.
* Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease must not require immediate CNS specific treatment at the time of study registration. Patients who have completed CNS therapy prior to starting therapy and clinically stabilized are also eligible.
* Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or make study participation not in the best interest of the patient, in the opinion of the treating investigator.
* Patient has known psychiatric or substance abuse disorders that, in the opinion of the investigator, would interfere with cooperation with the requirements of the trial.
* Pregnant patients or patients planning donation of sperm or breast milk during the therapy and for a minimum of 5 months after stopping therapy.
* Lactating patients if they do not agree to discontinue breast feeding through the entire duration of study participation and for 5 months after stopping therapy.
* History of another metastatic/relapsed active malignancy. Localized skin cancers such as basal cell or squamous cell cancer are allowed.
* Intractable nausea and vomiting refractory to therapy with antiemetics.
* History of hypersensitivity to ipilimumab, nivolumab, inulin or the formulations excipients.
* Known diagnosis of malabsorption disorder.
* Concurrent use of probiotics or antibiotics.
* Patients with a history of colectomy and/or gastric bypass.
* Patients with a known diagnosis of active inflammatory bowel disease or irritable bowel syndrome.
* History of organ transplant or stem cell/bone marrow transplant.
* Patients with active Clostridium difficile infection within 3 months before therapy start. Active infection is defined as a stool sample positive for Clostridium difficile toxin by enzyme immunoassay (EIA) and either symptoms (frequent loose stools) OR imaging findings consistent with toxic megacolon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2031-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression free survival (PFS) | At 6 months
  Will give an estimate and 95% confidence interval for the difference in the 6-month PFS rate between the combination arm and the single agent arm. This will be determined using binomial statistics. To allow for possible variability in the timing of the 6-month progression assessment, the 6-month PFS rate will be defined as the Kaplan-Meier estimate at 200 days after treatment initiation.
Incidence of inulin gel related adverse events | Up to 30 days after the last dose of inulin gel
  Will be reported descriptively. Toxicity will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

SECONDARY OUTCOMES:
Overall response rate | From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 3 years
  Will be assessed per Response Evaluation Criteria in Solid Tumors 1.1 criteria. An exact test for binomial proportion will be used. Will be assessed descriptively. Will be estimated with 95% confidence interval. Binomial statistics will be used for the binary outcomes.
Incidence of adverse events | Up to 30 days after the last dose of treatment
  Toxicity will be assessed according to the CTCAE, version 5.0.
PFS | From treatment start date to date of first documented disease relapse/progression, or death from cancer whichever occurs first, assessed up to 3 years
  Will be assessed descriptively. Will be estimated with 95% confidence intervals, for each treatment group separately. Kaplan-Meier plots for the time-to-event outcomes.
Overall survival | From treatment start date to death or last follow up, assessed up to 3 years
  Will be assessed descriptively. Will be estimated with 95% confidence intervals, for each treatment group separately. Kaplan-Meier plots for the time-to-event outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N Vaishampayan, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No